CLINICAL TRIAL: NCT00823706
Title: Prevalence of Chronic Angle Closure in Caucasian Hyperopic Subjects
Brief Title: Prevalence of Angle Closure in Caucasian Hyperopes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Yaniv Barkana, MD, Assaf-Harofeh Medical Center, Department of Ophthalmology
Other Study IDs: 122/08
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Angle Closure Glaucoma
Keywords: chronic angle closure hyperopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of this study is to assess the prevalence of asymptomatic chronic angle closure in high risk Caucasian individuals, namely those with hyperopia. A secondary purpose is to assess whether specific demographic or ocular-anatomic parameters in this population are associated with a higher risk for angle closure.

DETAILED DESCRIPTION:
Caucasian subjects aged > 40 years with hyperopia will undergo complete eye examination including subjective refraction and gonioscopy. In addition we will measure axial length, anterior chamber depth and lens thickness using ultrasound biometry.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 40 years
* Hyperopia greater then +1.00 D spherical equivalent

Exclusion Criteria:

* Any identifiable eye disease or previous eye surgery that can affect the anatomy of the irido-corneal angle

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caucasian subjects aged 40 years or more with hyperopia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-01

PRIMARY OUTCOMES:
prevalence of chronic angle closure in Caucasian hyperopes | 1 year

SECONDARY OUTCOMES:
relative risk for chronic angle closure measured for demographic and ocular-anatomic parameters | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofe Medical Center Ophthalmology Department, Ẕerifin, Israel